CLINICAL TRIAL: NCT04571541
Title: Outcomes of Endoscopic Management of Esophageal Wall Defects at a Large Referral Center
Brief Title: Endoscopic Management of Esophageal Wall Defects
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Mohammad Al-Haddad, Associate Professor of Medicine, Indiana University
Other Study IDs: 1509223988
Record Dates: First submitted 2020-09-26; First posted 2020-10-01 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Esophageal Fistula; Esophageal Perforation
MeSH Terms: conditions — Esophageal Fistula; Esophageal Perforation | interventions — Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Stenting — Effect of endoscopic stenting on healing of esophageal wall defects

SUMMARY:
The study aim at comparing outcomes from the implementation of various endoscopic closure techniques including stenting and suturing on the healing and resolution of esophageal wall defects.

DETAILED DESCRIPTION:
Esophageal wall defects are a rare but potentially life-threatening subset of luminal pathology which usually require timely intervention in order to reduce the known associated high morbidity and mortality. These defects can be due to surgical and endoscopic procedures, such as post-operative leaks and fistulas and perforations complicating endoscopic dilation. In addition, defects can occur spontaneously due to Boerhaave's syndrome or following chemoradiation treatments of esophageal or other chest malignancies. Surgical management was historically the mainstay of therapy for these defects with conservative management remaining an alternative in poor surgical candidates. Over the last several years however, interventional endoscopy has played an increasing role in treatment of esophageal wall defects, with endoscopic stenting quickly becoming a viable alternative. Temporary stents including the fully covered self-expandable metal stents (FC-SEMS), partially covered self-expandable metal stents (P-SEMS) and self-expandable plastic stents (SEPS) have all been successfully used and have become increasingly regarded as the new standard of care.

Indiana University is a tertiary referral center is a destination for complex thoracic surgery, oncology and esophageal disease referrals. The innovative luminal endoscopy team started employing a several modalities including flexible endoscopic suturing and stenting to close esophageal defects. To our knowledge, there is a dearth of data on outcomes associated with multi-modality esophageal defect closure techniques and little to no data comparing this approach to the current standard of care of stenting alone or surgery.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with spontaneous or iatrogenic esophageal wall defect

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients who present who our medical center with existing esophageal wall defect seeking endoscopic treatment and management
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Resolution of esophageal wall defect | 7/1/2014 to 7/1/2022
  Resolution of esophageal wall defect

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided